CLINICAL TRIAL: NCT00458653
Title: Vaccination With Dendritic Cell/Tumor Fusions in Conjunction With Autologous Stem Cell Transplant in Patients With Multiple Myeloma
Brief Title: Vaccination With Dendritic Cell/Tumor Fusions With Autologous Stem Cell Transplants in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Massachusetts General Hospital (Other); Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, David Avigan, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-098
Record Dates: First submitted 2007-04-10; First posted 2007-04-11 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma
Keywords: DC/tumor cell fusions; GM-CSF; high dose chemotherapy
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Post-transplant vaccination
  Interventions: Biological: Dendritic Cell Tumor Fusion
- Group B (Experimental): Pre- and post-transplant vaccination
  Interventions: Biological: Dendritic Cell Tumor Fusion

INTERVENTIONS:
Biological: Dendritic Cell Tumor Fusion — Post-Transplant (Groups A and B): Given under the skin every four weeks for three doses.
  Pre-Transplant (Group B): Injected under the skin in upper part of leg or arm prior to stem cell collection for ASCT

SUMMARY:
The main purpose of this study is to test the safety and determine the type and severity of any side effects of the Dendritic Cell Fusion Vaccine given in combination with an autologous transplant for patients with multiple myeloma. Autologous stem cell transplantation is a standard therapy for multiple myeloma that is often successful in significantly decreasing the amount of cancer. However, it is not a cure because at some point the multiple myeloma generally begins to grow again. Cancer vaccines are investigational agents that try to stimulate the immune system to recognize and fight against cancer cells. One type of cancer vaccine uses an immune stimulating cell of the body known as a dendritic cell. Research has shown that these dendritic cells can stimulate an immune response against the tumor.

DETAILED DESCRIPTION:
* The first group of participants on this study will receive up to 3 monthly doses of the study vaccine beginning about 1 month following the autologous transplant. If this is found to be safe, the next group will receive one additional study vaccine prior to the transplant and then up to 3 doses after the transplant.
* If the screening tests determine that the participant is eligible for the study, they will undergo dendritic cell collection by a procedure called leukapheresis. Leukapheresis involves the collection of white blood cells from the blood. Dendritic cells are grown from these white blood cells in the laboratory. Tumor cells will also be collected from the bone marrow through a bone marrow aspirate/biopsy.
* After cells have been collected for study vaccine generation, the participant may receive standard therapy to reduce the number of multiple myeloma cells in the body. The specific regimen will be determined by the participants multiple myeloma physician.
* The first group of patients will receive the study vaccine only after the transplant. If this is found safe then the second group will receive a single study vaccine prior to the transplant.
* Prior to the autologous stem cell transplant, we will harvest stem cells from the participants blood that will be used for the transplant later. G-CSF will be given as a daily injection beginning the day after the chemotherapy and GM-CSF injections will be started seven days after the chemotherapy. These injections will continue until after the stem cells are collected. Approximately 10 days after the chemotherapy, participants will undergo a leukapheresis procedure to collect the stem cells.
* Within a few weeks of successful stem cell collection, the participant will be admitted to the hospital for high dose chemotherapy with autologous stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma who are potential candidates for high dose chemotherapy
* Measurable disease as defined by a history of an elevated M component in plasma, urine, or free kappa/lambda light chains in the serum
* 18 years of age or older
* ECOG Performance Status of 0-1 with greater than a nine week life expectancy
* Patients with > 20% bone marrow involvement or plasmacytoma amenable to resection under local anesthesia
* Negative pregnancy test, and adequate contraception method
* DLCO (adjusted)> 50%
* Cardiac Ejection Fraction > 45%
* Laboratory values within the ranges outlined in the protocol

Exclusion Criteria:

* History of clinically significant venous thromboembolism
* Clinically significant autoimmune disease
* HIV positive
* Serious intercurrent illness such as infection requiring IV antibiotics, or significant cardiac disease characterized by significant arrhythmia, ischemic coronary disease or congestive heart failure
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-04; Primary Completion 2012-04 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
To assess the toxicity associated with vaccination of multiple myeloma patients with dendritic cell/myeloma fusions and GM-CSF prior to stem cell mobilization and following high dose chemotherapy with stem cell rescue. | 5 years

SECONDARY OUTCOMES:
To determine whether tumor specific cellular and humoral immunity can be induced by serial vaccination with DC/tumor cell fusions in conjunction with high dose chemotherapy with stem cell rescue | 5 years
To determine if vaccination with DC/tumor cell fusions results in clinical disease response in patients with evidence of residual disease post-transplant | 5 years
To determine the time to disease progression in this participant population.

CONTACTS AND LOCATIONS:
Overall Officials: David Avigan, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (4):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute/Brigham & Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
- Rambam Medical Center, Haifa, Israel